CLINICAL TRIAL: NCT03247322
Title: Improving Transplant Medication Safety Through A Pharmacist-Empowered, Patient-Centered, Mhealth-Based Intervention (TRANSAFE Rx Study)
Brief Title: mHealth Medication Safety Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00068746
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Medication Compliance
Keywords: Medication Safety; Mobile Health Technology
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In order to minimize bias, data for outcomes will be collected by a blinded study coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Group (Experimental): Patients in the intervention cohort will have enhanced medication safety monitoring utilizing a Pharmacist-led medication therapy using mHealth application. The application will provide patients a useful tool to conduct self-care monitoring and management, including timely reminders to take medications, automated messages when patients miss multiple medication doses, tracking of medication side effects and reporting trends in blood pressures and glucoses (when applicable).
  Interventions: Other: Pharmacist-led medication therapy using mHealth application
- Usual Care Group (No Intervention): Subjects in the control group will receive the usual standard of follow up care for kidney transplant patients.

INTERVENTIONS:
Other: Pharmacist-led medication therapy using mHealth application — This cohort of participants will receive clinical pharmacist-led supplemental medication therapy monitoring and management, utilizing a smartphone-enabled mHealth application, integrated with televisits and home-based monitoring of blood pressures and glucoses (when applicable).
  Arms: mHealth Group

SUMMARY:
TRANSAFE Rx is a 12-month, parallel two-arm, 1:1 randomized controlled clinical trial, involving 136 participants (68 in each arm) measuring the clinical and economic effectiveness of a pharmacist-led intervention, which utilizes an innovative mHealth application to improve medication safety and health outcomes, as compared to usual post-transplant care. The primary goal of the TRANSAFE Rx study is to demonstrate significant reductions in med safety issues leading to reduced healthcare resource utilization in kidney transplantation through a pharmacist-led, mHealth-enabled, intervention. This study will provide detailed and novel information on the incidence, etiologies and outcomes of med errors and adverse drug events in this high-risk population; while also demonstrating the effectiveness of this intervention on reducing the incidence and impact of med safety issues in kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient between 6 and 36 months post-transplant
* At least 18 years of age
* Transplant MD agrees that patient is eligible to participate

Exclusion Criteria:

* Multi-organ recipient
* Patient is incapable of:
* Measuring their own blood pressure and glucose (if applicable)
* Self-administering medications
* Speaking, hearing and reading English
* Utilizing the mHealth application, after training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Taber, PharmD,MS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Gonzales HM, Fleming JN, Gebregziabher M, Posadas Salas MA, McGillicuddy JW, Taber DJ. A Critical Analysis of the Specific Pharmacist Interventions and Risk Assessments During the 12-Month TRANSAFE Rx Randomized Controlled Trial. Ann Pharmacother. 2022 Jun;56(6):685-690. doi: 10.1177/10600280211044792. Epub 2021 Sep 8. PMID 34496669
- [Derived] Taber DJ, Fleming JN, Su Z, Mauldin P, McGillicuddy JW, Posadas A, Gebregziabher M. Significant hospitalization cost savings to the payer with a pharmacist-led mobile health intervention to improve medication safety in kidney transplant recipients. Am J Transplant. 2021 Oct;21(10):3428-3435. doi: 10.1111/ajt.16737. Epub 2021 Jul 14. PMID 34197699
- [Derived] Fleming JN, Treiber F, McGillicuddy J, Gebregziabher M, Taber DJ. Improving Transplant Medication Safety Through a Pharmacist-Empowered, Patient-Centered, mHealth-Based Intervention: TRANSAFE Rx Study Protocol. JMIR Res Protoc. 2018 Mar 2;7(3):e59. doi: 10.2196/resprot.9078. PMID 29500161

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | mHealth Group | Usual Care Group
Started | 68 | 68
Completed | 66 | 68
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Patients in the intervention cohort will have enhanced medication safety monitoring utilizing a Pharmacist-led medication therapy using mHealth application. The application will provide patients a useful tool to conduct self-care monitoring and management, including timely reminders to take medications, automated messages when patients miss multiple medication doses, tracking of medication side effects and reporting trends in blood pressures and glucoses (when applicable).
  Pharmacist-led medication therapy using mHealth application: This cohort of participants will receive clinical pharmacist-led supplemental medication therapy monitoring and management, utilizing a smartphone-enabled mHealth application, integrated with televisits and home-based monitoring of blood pressures and glucoses (when applicable).
- Control Group: Subjects in the control group will receive the usual standard of follow up care for kidney transplant patients.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 51 (14) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 35 | 42 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 19 | 46
  Black | 40 | 47 | 87
  Hispanic | 1 | 2 | 3
Number of Participants with History of Diabetes [Count of Participants; unit: Participants] | 19 | 35 | 54
Number of Participants with History of Hypertension [Count of Participants; unit: Participants] | 63 | 61 | 124
Number of Participants on Dialysis at Transplant [Count of Participants; unit: Participants] | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Medication Errors
Description: Medication errors will be defined as documentation that a patient is taking a medication in a manner that was not intended
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: number of medication errors
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 68 | 68
number of medication errors | 9 (5.4) | 20 (14)

2. Primary Outcome: Incidence and Severity of Adverse Drug Events
Description: Adverse Events will be defined according to the AHRQ Patient Safety Network as an injury resulting from medical care.
  Rates of Events Per Patient Year by AE Grade
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: adverse events per patient year
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 68 | 68
adverse events per patient year
  Overall | 20.68 (18.35) | 21.26 (25.24)
  Grade 1 | 13.96 (1.47) | 14 (15.10)
  Grade 2 | 5.53 (0.72) | 5.28 (0.94)
  Grade 3 | 1.10 (.22) | 1.57 (.34)
  Grade 4 | .07 (.05) | 0.38 (.15)
  Grade 5 | 0 (0) | .01 (.01)
  Grade 3 or higher | 1.18 (.25) | 1.97 (.46)

3. Primary Outcome: Severity of Medication Errors
Description: Severity of Medication Errors were measured using the Overhage criteria
Time Frame: 1 year
Measure: Number; unit: number of medication errors
Arm/Group | mHealth Group | Usual Care Group
Number analyzed (Participants) | 68 | 68
number of medication errors
  Potentially Lethal | 0 | 0
  Serious | 0 | 1
  Significant | 586 | 1320
  Minor | 28 | 64

4. Secondary Outcome: Hospitalization Rate
Description: Number of hospitalizations per patient-year
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Hospitalizations per patient-year
Arm/Group | mHealth Group | Usual Care Group
Number analyzed (Participants) | 68 | 68
Hospitalizations per patient-year | 0.65 [0.4 to 0.94] | 1.08 [0.60 to 1.6]

5. Other Pre Specified Outcome: Infection Rate
Description: Number of infections per patient-year
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Infections per patient-year
Arm/Group | mHealth Group | Usual Care Group
Number analyzed (Participants) | 68 | 68
Infections per patient-year | 1.32 [0.92 to 1.72] | 1.26 [0.76 to 1.76]

6. Other Pre Specified Outcome: Opportunistic Infection Rate
Description: Opportunistic infections per patient-year
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Opportunistic infection per patient-year
Arm/Group | mHealth Group | Usual Care Group
Number analyzed (Participants) | 68 | 68
Opportunistic infection per patient-year | .19 [.09 to 0.30] | .14 [.01 to .30]

ADVERSE EVENTS:
Time Frame: 1 year
Description: The data was analyzed by adverse event type and severity, not specific adverse event terms.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 6/68 | 16/68
Other Adverse Events (participants affected / at risk) | 68/68 | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=68) | Control Group (N=68)
GI Dysfunction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Laboratory abnormality (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
General Disorder (General disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 3 (3)
Psychiatric Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Abnormal Vital Signs (General disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=68) | Control Group (N=68)
Hypertension (Cardiac disorders) | 59 (59) | 63 (63)
Ear disorders (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 30 (30) | 29 (29)
Procedural complications (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Laboratory Abnormality (Investigations) | 64 (64) | 64 (64)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10)
Nervous System Disorder (Nervous system disorders) | 23 (23) | 19 (19)
Psychiatric Disorders (Psychiatric disorders) | 4 (4) | 5 (5)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 7 (7)
Skin disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03247322/Prot_SAP_000.pdf